CLINICAL TRIAL: NCT06116877
Title: Effect of Adding Zirconium Oxide Nanoparticles to Printable Implant Overdenture Acrylic Resin Base Material. Clinical Comparative Study
Brief Title: Effect of Adding Zirconium Oxide Nanoparticles to Printable Implant Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A03010322
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (I) non modified (Active Comparator): Five patients will receive mandibular 2-implant retained overdentures of non-modified printable acrylic resin base material.
  Interventions: Procedure: implant supported overdenture
- Group (II) modified (Active Comparator): Five patients will receive mandibular 2-implant retained overdentures of modified printable acrylate resin base material with zirconium oxide nanoparticles.
  Interventions: Procedure: implant supported overdenture

INTERVENTIONS:
Procedure: implant supported overdenture — mandibular 2-implant retained overdenture of non-modified printable acrylate resins base material with Zirconium oxide nanoparticles

SUMMARY:
This clinical study will be conducted to evaluate and compare non-modified printable acrylic resin base material and modified printable acrylic resin base material with zirconia oxide nanoparticles for a 2-implant retained complete overdenture regarding:Surface roughness; microbiological assessment of denture base microbiological analysis peri-implant soft tissue health around used implants

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients are healthy, free from any systemic diseases relating to bone resorption such as uncontrolled diabetics or osteoporosis. This will be achieved through medical history and clinical examination by physician.

  2. They will have completely edentulous jaws for at least 1 year. 3. They will be of angle's class I maxillo-mandibular relationship and have upper and lower completely edentulous arches.

  4. Residual alveolar ridges covered with healthy firm mucosa. 5. All included patients will have sufficient available length and width of mandibular bone to accommodate conventional implant. (At least 5 mm buccolingual width and 12 mm vertical height of bone.

Exclusion Criteria:

* Patients with chronic systemic diseases that affect bone metabolism
* Uncontrolled diabetic patients
* Patients with TMJ dysfunction
* Smokers

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Surface roughness | one year
  Surface roughness: will be evaluated using profilometer device
Microbiological assessment | one year
  Microbiological assessment of denture base surface microbiological analysis
Peri-implant soft tissue health | one year
  was evaluated using scores for plaque and gingival bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University ,Faculty of dentistry, Al Mansurah, Egypt